CLINICAL TRIAL: NCT02713880
Title: Biomarker for Transthyretin-Related Familial Amyloidotic Polyneuropathy - An International, Multicenter, Epidemiological Protocol
Brief Title: Biomarker for Transthyretin-Related Familial Amyloidotic Polyneuropathy (BioTRAP)
Acronym: BioTRAP
Status: Withdrawn | Type: Observational
Why Stopped: University of Rostock terminated participation in the study conduct; Study Sponsorship is moved to Centogene AG
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BTR 06-2018
Record Dates: First submitted 2016-01-13; First posted 2016-03-21 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Transthyretin Amyloidosis; Transthyretin-Related (ATTR) Familial Amyloid Polyneuropathy; Transthyretin Amyloid Cardiopathy
Keywords: Amyloid Neuropathies; Biomarker
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Amyloid Neuropathies, Familial; Amyloid Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectometry, maximal 7,5 blood will be taken from the patient via a dry blood spot filter card. To proof the correct diagnosis in those patients where up to the enrolment in the study no genetic testing has been done, sequencing will be done. The analyses will be done at the Centogene GmbH Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Transthyretin-Related Familial: Patients with Transthyretin-Related Familial Amyloidotic Polyneuropathy or high-grade suspicion for Transthyretin-Related Familial Amyloidotic Polyneuropathy

SUMMARY:
International, multicenter, observational, longitudinal study to identify biomarker/s for the development of a new MS-based biomarker for the early and sensitive diagnosis of Transthyretin-Related Familial Amyloidotic Polyneuropathy from blood and number of correctly identified patients with Transthyretin-Related Familial Amyloidotic Polyneuropathy

DETAILED DESCRIPTION:
Diseases of diverse etiology can be correlated to the term "polyneuropathy"(PNP). The pathogenesis may be of inflammatory, autoimmune, metabolic, toxic or hereditary nature. Careful clinical and electrodiagnostic assessment, with attention to the pattern of involvement and the types of nerve fibers most affected, narrows the differential diagnosis and helps to focus the laboratory evaluation. Beside the frequent genetic etiologies in PNP (pmp22, MFN2) one cause of a polyneuropathy may be a hereditary amyloidosis. This term describes the accumulation of misfolded protein in the interstitial space. The abnormal accumulation of β-fibrils can be detected histologically by Congo pink staining. Aside from acquired amyloidotic neuropathies (e.g. PNP caused by AL-amyloidosis [AL= amyloidosis with light chain immunoglobins]) there are also hereditary amyloidotic neuropathies.

These have been described as endemic in Sweden, Portugal or Japan. More recent studies provided evidence for the presence of hereditary amyloidotic neuropathies amongst the German population and that they are currently underdiagnosed. The most common form of the hereditary familial amyloidotic neuropathy (FAP) is the Transthyretin-related FAP, however two other amyloidogenic proteins have been described: Apolipoprotein A-I and Gelsolin (Ando et al., 2005; Adams et al., 2010).

The TTR-FAP is an autosomal dominant disease, the exact prevalence of which is unknown but estimated to be around 1:100,000 to 1:1,000,000 in the normal population. By limiting the study population to patients with PNP of unknown etiology it should be possible to gain evidence for the prevalence of the disease in Germany by investigating fewer patients.

While the diagnosis of the amyloidotic neuropathy can be conducted histologically, a molecular genetic approach is necessary to diagnose TTR-FAP. Even though more than 100 point mutations are known to cause the disease, the most common amino acid change is V30M.

The mutation in the TTR gene causes the destabilization of the physiologically tetrameric protein. Usually transthyretin consists of four identical monomeric subunits and binds the thyroxin circulating in the blood plasma. The monomeric subunits exhibit a pronounced β- sheet structure which leads to the accumulation of unsoluble β-fibrils when they are destabilised as in TTR-FAP.

This accumulation of misfolded TTR can lead to three phenotypes known as:

* cardiac TTR amyloidosis
* leptomeningeal TTR amyloidosis and the
* TTR-FAP

The TTR-FAP has a very heterogeneous phenotype which can manifest starting at the age of 18 and may lead to death within 10 years. The symptoms can be categorized in three groups (Ando et al. 2005):

Dysfunction of peripheral nerves:

* Dissociated anesthesia
* Muscle paresis and atrophy
* Dysaesthesia and paraesthesia
* Reduced skin temperature
* Coldness
* Hoarseness

Autonomic dysfunction:

* Dysuria
* Diarrhea
* Constipation
* Orthostatic dysregulation
* Erectile dysfunction
* Nausea

Constitutional conditions

* Anemia
* Weight loss
* Arrhythmia
* Edema
* Acroparaesthesia

The currently available therapeutic approaches are either liver transplantation (as the liver mainly produces transthyretin this is a feasible approach) or as of more recently also a TTR- tetramer stabilizing agent (Tafamidis). Tafamidis (Vyndaqel®) gained the European approval under "exceptional circumstances"in November 2011 for treating FAP in adults with a symptomatic polyneuropathy. In light of the potential therapy of this very rare disease, this study aims to determine the prevalence of TTR-FAP in a selected, clinical subpopulation. New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood (plasma) of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the plasma of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained from the parents before any study related procedures.
* Patients of both genders older than 2 months
* The patient has a diagnosis of Transthyretin-Related Familial Amyloidotic Polyneuropathy or a high-grade suspicion for Transthyretin-Related Familial Amyloidotic Polyneuropathy
* High-grade suspicion present, if one or more inclusion criteria are valid:

  * Positive family anamnesis for Transthyretin-Related Familial Amyloidotic -Polyneuropathy
  * Orthostatic dysregulation
  * Acroparaesthesia
  * Dysaesthesia and paraesthesia
  * Muscle paresis and atrophy

Exclusion Criteria:

* No Informed consent from the parents before any study related procedures.
* Patients of both genders younger than 2 months
* No diagnosis of Transthyretin-Related Familial Amyloidotic Polyneuropathy or no valid criteria for profound suspicion of Transthyretin-Related Familial Amyloidotic Polyneuropathy

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Transthyretin-Related Familial Amyloidotic Polyneuropathy or high-grade suspicion for Transthyretin-Related Familial Amyloidotic Polyneuropathy
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Transthyretin-Related Familial Amyloidotic Polyneuropathy from blood | 36 months

SECONDARY OUTCOMES:
Number of correctly identified patients with Transthyretin-Related Familial Amyloidotic Polyneuropathy | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Rolfs, Prof., Principal Investigator — CENTOGENE GmbH Rostock
Locations (2):
- Centogene GmbH, Rostock, Germany
- Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai, India

IPD SHARING:
Plan to Share IPD: Undecided